CLINICAL TRIAL: NCT01150240
Title: Clinical and Laboratory Online Patient- and Research Database for Primary Immunodeficiencies in Switzerland
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Collaborators: University of Basel (Other); University of Bern (Other); University Hospital, Geneva (Other); University of Lausanne (Other); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Other Study IDs: PID_CH_Registry06
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Primary Immunodeficiency Disease
Keywords: Primary Immunodeficiency Disease
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (1):
- Primary Immunodeficiency Disease: Patients with primary Immunodeficiency disease (PID)

SUMMARY:
A Swiss national, multi-centre, online patient and research database will be created, using the existing ESID database server system. This database contains disease-specific data from patients with primary (inborn) immunodeficiency diseases (PID).

DETAILED DESCRIPTION:
The project aims to compile clinical and laboratory data of patients with primary immunodeficiencies (PID) in order to improve diagnosis, classification, prognosis and therapy. The online technology offers features not available in former databases such as access control,security functionality, and maintenance of data integrity during transactions and system errors, online back up, online optimization, scalability and online SQL-queries as well as a long term documentation of patients.

Furthermore the database can be used for the submission and storage of molecular diagnostic results and thus allow the compilation of genotype and phenotype observations, which is of essential and immediate use for the patient himself and patient care. An attending physician may gain information on similar cases of a rare PID disease in Switzerland and European countries and use these insights for therapy. In addition, it will be possible to obtain an insight on side effects. Thus, the system also meets the requirements of an optimal platform for Phase IV studies of post-licensing drug surveillance-programs.

ELIGIBILITY:
Inclusion Criteria:

* Primary Immunodeficiency Disease (PID)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Primary Immunodeficiency Disease (PID), followed in a PID centre, primary care hospitals or private practice
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2006-10; Primary Completion 2018-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Helbling, Prof., Principal Investigator — University Bern, Inselspital; Christoph Hess, Prof., Principal Investigator — University Basel, University Hospital; Ayse H Ozsahin, Prof., Principal Investigator — University Geneva, University Hospital; Francois Spertini, Prof., Principal Investigator — University Lausanne, University Hospital; Hugo Ubieto, MD, Principal Investigator — Department of Child Development, Children's Hospital St. Gallen, Switzerland; Reinhard A Seger, Prof., Principal Investigator — University Zürich, University Children's Hospital
Locations (6):
- Switzerland (6):
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern
  - University Children's Hospital Geneva, Geneva
  - University Hospital Lausanne, Lausanne
  - Children's Hospital of Eastern Switzerland and Cantonal Hospital, Sankt Gallen
  - University Children's Hospital Zurich, Zurich